CLINICAL TRIAL: NCT01412788
Title: Randomized Controlled Trial of Safety and Aesthetic Outcomes of Breast-conserving Surgery With the Peri-areolar Incision Approach
Brief Title: Safety and Aesthetic Outcomes of Breast Conserving Surgery With Peri-areolar Incision Approach
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Qiang Sun, the department of breast surgery of PUMCH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH- BCS
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; Breast Conserving Surgery; Peri-areolar Incision
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peri-areolar incision (Experimental): Peri-areolar incision was used to carry out lumpectomy
  Interventions: Procedure: peri-areolar incision
- traditional incision (Active Comparator): traditional incision above tumor was used to carry out lumpectomy
  Interventions: Procedure: traditional incision

INTERVENTIONS:
Procedure: peri-areolar incision — peri-areolar incision was used to carry out lumpectomy in breast-conserving surgery.
  Arms: peri-areolar incision
Procedure: traditional incision — Traditional incision above tumor was used to carry out breast-conserving surgery.
  Arms: traditional incision

SUMMARY:
Cosmetic result after breast-conserving surgery (BCS) would impose great effect upon patient's quality of life. Although peri-areolar incision has been widely used in benign breast tumor excision, mastopexy procedures and skin-sparing mastectomy with primary reconstruction, the actual safety and aesthetic outcome of the peri-areolar incision approach in BCS for cancer patients has not been established by randomized, controlled trials.

This trial was design to compare the Safety and aesthetic outcomes of breast conserving surgery between peri-areolar incision approach and traditional methods.

DETAILED DESCRIPTION:
The Trial aims to determine whether BCS with the peri-areolar approach: 1) is safe in terms of the rates of recurrence and metastasis; 2) can improve the post-operative aesthetic score and QOL score.

ELIGIBILITY:
Inclusion Criteria:

* patients desire for breast conserving surgery;
* fulfills criteria for breast conserving surgery;
* the maximum diameter of the tumor should be less than the semi-perimeter of the areola and that the proximal margin of tumor should be at least 1 cm away from the areola;
* patients suitable to receive BCS with either the peri-areolar incision or the traditional incision were included;

Exclusion Criteria:

* patients not suitable for breast conserving surgery;
* skin or sub-cutaneous tumor invasion as definite contra-indication of skin-sparing;
* male or bilateral breast cancers who might bring up bias in deciding aesthetic outcomes and expenditure;
* Patients who were supposed to benefit from a certain kind of incision were also excluded at the researcher's discretion.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
event free survival | 5 years
  local recurrence, regional recurrence, distant metastasis, death

SECONDARY OUTCOMES:
aesthetic outcomes | two weeks, half a year and one year
  aesthetic score and QOL score
cost | 2 weeks
  operation time for the surgery, hospital stay days, costs

CONTACTS AND LOCATIONS:
Overall Officials: Sun Qiang, Master, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China